CLINICAL TRIAL: NCT05161559
Title: Adhesive Performance of Glass Ionomer Versus Resin Based Adhesive Systems
Brief Title: Adhesive Performance of Glass Ionomer and Resin Based Adhesive Systems: A 3 Years Prospective Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A12151221
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Dental Leakage
Keywords: Resin Composite; Randomized Clinical Trial; Operative Dentistry
MeSH Terms: conditions — Dental Leakage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fuji Bond LC (Glass ionomer based adhesive) (Experimental): Patients received in Class V cavity preparation Fuji Bond LC (Glass ionomer based adhesive) on one tooth of the mouth
  Interventions: Procedure: Chemical bond adhesive (GC, Corporation, Tokyo, Japan)
- Riva Bond LC (Glass ionomer based adhesive) (Experimental): Patients received in Class V cavity preparation Riva Bond LC (Glass ionomer based adhesive) on one tooth of the mouth
  Interventions: Procedure: Chemical bond adhesive (GC, Corporation, Tokyo, Japan)
- Single Bond Universal (self-etch adhesive) (Experimental): Patients received in Class V cavity preparation Single Bond Universal (self-etch adhesive) on one tooth of the mouth
  Interventions: Procedure: Self-etch adhesive (Kuraray, Tokyo, Japan)
- Clearfill S3 Bond (self-etch adhesive) (Experimental): Patients received in Class V cavity preparation Clearfill S3 Bond (self-etch adhesive) on one tooth of the mouth
  Interventions: Procedure: Self-etch adhesive (Kuraray, Tokyo, Japan)
- OptiBond FL (three step etch & rinse adhesive) (Experimental): Patients received in Class V cavity preparation OptiBond FL (three step etch & rinse adhesive) on one tooth of the mouth
  Interventions: Procedure: Etching with phosphoric acid gel (3M ESPE, St. Paul, MN, USA)

INTERVENTIONS:
Procedure: Etching with phosphoric acid gel (3M ESPE, St. Paul, MN, USA) — Etching enamel surface using phosphoric acid gel (3M ESPE, St. Paul, MN, USA)
  Arms: OptiBond FL (three step etch & rinse adhesive)
Procedure: Self-etch adhesive (Kuraray, Tokyo, Japan) — No Etching enamel surface using phosphoric acid (self-etch technique) (Kuraray, Tokyo, Japan)
  Arms: Clearfill S3 Bond (self-etch adhesive); Single Bond Universal (self-etch adhesive)
Procedure: Chemical bond adhesive (GC, Corporation, Tokyo, Japan) — Chemical bond with hydroxyapatite crystals of Enamel (GC, Corporation, Tokyo, Japan)
  Arms: Fuji Bond LC (Glass ionomer based adhesive); Riva Bond LC (Glass ionomer based adhesive)

SUMMARY:
This study aimed to clinically evaluate the 3-years clinical performance of glass ionomer and resin based adhesive systems in Class V restorations.

DETAILED DESCRIPTION:
The formulated null hypothesis was that there is no significant difference in the clinical performances between glass ionomer and resin based adhesive systems in Class V restorations for 3-years.

The research question was as follows: Do glass ionomer adhesives in class V restorations present better clinical performances than resin based adhesive systems according to the modified United States Public Health Service (modified-USPHS) criteria?

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary caries involving cervical surface only with ICDAS 2 and 3.
2. Patients with normal and full occlusion.
3. Patients with tooth gives positive response to testing with an electric pulp tester.
4. Patients must have a good oral hygiene.
5. Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

1. High caries risk patients with extremely poor oral hygiene.
2. Patients involved in orthodontic treatment or periodontal surgery.
3. Patients with periodontally involved teeth (chronic periodontitis).
4. Patients with heavy bruxism habits and clenching.
5. Patients with abutments should be excluded.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage % of patients with marginal staining | 3 years after restoration procedure
  Percentage of marginal staining in patients was clinically assessed using USPHS criteria. Restorations were given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study Protocol, Statistical Analysis Plan can be shared to other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 3 Months for 5 years
Access Criteria: For anyone